CLINICAL TRIAL: NCT05899413
Title: Examining Transcutaneous Vagal Nerve Stimulation as a Facilitator of Social Bonding
Acronym: CtVNS
Status: Completed | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 23-39189; U24AG072699 (NIH)
Record Dates: First submitted 2023-05-24; First posted 2023-06-12 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Vagus Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Couple dyads will be randomly assigned to receive either tVNS or sham stimulation.
Who Masked: Participant
Masking Description: Participant couples will be blinded to their condition. Experimenters running the study will not be blinded since tVNS administration currently requires their knowledge of the condition.
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Active tVNS (Experimental): We will use a research edition of an auricular vagus nerve stimulator (tVNS RE, Vagus.net™, UK) that sends current-controlled stimulation in symmetric biphasic waveforms. The tVNS RE conforms to EU directive 93/42/EEC medical device standards and ISO/IEC 17050-1. This device consists of a handheld stimulator and an electrode clip. We will deliver stimulation at the individually calibrated intensity continuously during the interactions, and the default device settings we adopted were as follows: frequency = 30Hz, phase duration = 250μs, interphase interval = 50μs, and max voltage = 65V. In the active stimulation condition, both partners will have the stimulation clip attached to the outer auditory canal.
  Interventions: Device: Transcutaneous vagal nerve stimulation
- Sham tVNS (Sham Comparator): In the sham condition, both partners will have electrodes attached to the center of the left ear lobe. They will still receive stimulation but at a placement that should not activate the vagus nerve.
  Interventions: Device: Transcutaneous vagal nerve stimulation

INTERVENTIONS:
Device: Transcutaneous vagal nerve stimulation — The intervention consists of neurostimulation device that is programmed to a stimulus intensity at 0.5mA with a stimulation frequency of 25 Hz at the outer auditory canal.

SUMMARY:
This study aims to understand the role of the vagus nerve in promoting social bonding by using a non-invasive stimulation technique called transcutaneous vagal nerve stimulation (tVNS). The investigators will investigate whether tVNS can improve emotional, physiological, and behavioral experiences during and after social interactions. Couples will be randomly assigned to receive either tVNS or a sham stimulation during gratitude expression and problem-solving discussions. The investigators will measure their subjective evaluations of the interactions and capture their physiological and behavioral synchrony. This research will shed light on the processes involved in social connection and explore the potential of tVNS as a tool to enhance bonding in close relationships.

DETAILED DESCRIPTION:
As fundamental as the need to belong is to human survival and functioning, decades of research have shown that social connection is critical to emotional well-being. The current investigation seeks to use the knowledge and technological advances in the biomedical field to examine the causal role of the vagus nerve in promoting social bonding. Specifically, building on the recent evidence suggesting the effects of transcutaneous vagal nerve stimulation (tVNS) on improving social cognitive functioning, this study will examine the utility of tVNS in modulating emotional, physiological, and behavioral experiences during and after social interactions. The investigators will examine if romantic couple assigned to receive tVNS vs. active sham stimulation during two types of conversations (i.e., gratitude expression and problem-solving discussion) show differences in their experiences of the interactions. The study outcomes will include subjective evaluations of the interaction (e.g., felt emotions) and their physiological synchrony. This investigation will provide insights into the mechanistic processes that undergird social connection and, importantly, be the first to examine the potential utility of tVNS as an intervention tool for promoting social bonding within close relationships.

ELIGIBILITY:
Inclusion Criteria:

* Fluent in English
* Having been in a relationship with the partner for at least a year
* Within the age range of 18-39

Exclusion Criteria:

* Major chronic disease. self-reported autoimmune disease; severe asthma; lung disease (such as chronic bronchitis; history of stroke, heart attack, epilepsy, brain injury); cardiovascular disease.
* Cancer: if not in remission.
* Substance dependence-current or long history (5 years of more).
* Current psychiatric diagnosis that is not being treated with medication
* Confounding medications, including those used to treat hypertension and cardiovascular conditions; psychoactive substances; and medications known to directly affect autonomic functioning.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Nancy Friend Pritzker Psychiatry Building, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
There is currently no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Chung JM, Harari GM, Denissen JJ. Investigating the within-person structure and correlates of emotional experiences in everyday life using an emotion family approach. Journal of Personality and Social Psychology. 2022;122(6):1146-1189.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 80 couples (i.e., 160 participants) were recruited from February 2024.
Pre-assignment Details: Couples were randomly assigned to either the active or sham stimulation condition after confirming their eligibility and completing a background questionnaire at home. Although all sessions were completed, technical issues (e.g., tVNS device malfunction) occurred in some cases. When this happened, the affected couple was excluded from the random assignment, and the next couple was reassigned to that condition.
Groups:
- Active tVNS: We delivered stimulation at the individually calibrated intensity continuously during the interactions, and the default device settings we adopted were as follows: frequency = 30Hz, phase duration = 250μs, interphase interval = 50μs, and max voltage = 65V. In the active stimulation condition, both partners will have the stimulation clip attached to the outer auditory canal. In the sham stimulation condition, they will have the stimulation clip attached to their earlobe.
Period: Overall Study
Arm/Group | Active tVNS | Sham tVNS
Started | 86 | 74
Completed | 86 | 74
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: After excluding five individuals whose physiological data during the conflict were unavailable and one whose baseline RSA was unavailable, our final analytic sample consisted of 134 individuals.
Groups:
- Active tVNS: We delivered stimulation at the individually calibrated intensity continuously during the interactions, and the default device settings we adopted were as follows: frequency = 30Hz, phase duration = 250μs, interphase interval = 50μs, and max voltage = 65V. In the active stimulation condition, both partners will have the stimulation clip attached to the outer auditory canal.
- Total: Total of all reporting groups
Arm/Group | Active tVNS | Sham tVNS | Total
Number analyzed (Participants) | 63 | 71 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.17 (4.33) | 27.65 (4.26) | 27.90 (4.29)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female/Male/Other: Female | 30 | 34 | 64
  Female/Male/Other: Male | 32 | 34 | 66
  Female/Male/Other: Other | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 27 | 35 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 33 | 23 | 56
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 1 | 4 | 5
Relationship duration [Mean (Standard Deviation); unit: Years] — how long the couple has been together in years
  Years | 4.23 (3.06) | 4.41 (2.41) | 4.33 (2.73)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Positive Affect
Description: During the conversation, overall, I felt… (1: not at all positive, 7: extremely positive)
Time Frame: Once, self-reported in a survey immediately following conflict interaction, up to 10 minutes
Population: Our analysis included 134 participants with complete physiological and self-report data. Missing data resulted from session failures (e.g., unstable or missing physiological measurements) or survey non-response
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tVNS | Sham tVNS
Number analyzed (Participants) | 63 | 71
units on a scale | 5.89 (0.92) | 5.69 (1.15)

2. Primary Outcome: Self-reported Negative Affect
Description: During the conversation, overall, I felt… (1: not at all negative, 7: extremely negative)
Time Frame: Once, self-reported in a survey immediately following conflict interaction, up to 10 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Active tVNS | Sham tVNS
Number analyzed (Participants) | 63 | 71
units on a scale | 5.79 (1.18) | 5.62 (1.32)

3. Primary Outcome: Respiratory Sinus Arrhythmia
Description: RSA was assessed continuously throughout the conversation.
Time Frame: Continuously throughout conflict conversation
Population: as for outcome 1
Measure: Mean (Standard Error); unit: ms
Arm/Group | Active tVNS | Sham tVNS
Number analyzed (Participants) | 63 | 71
ms | 6.47 (0.74) | 6.54 (0.89)

4. Primary Outcome: Interbeat Interval
Description: IBI was assessed continuously throughout the conversation.
Time Frame: Continuously throughout the conflict conversation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Active tVNS | Sham tVNS
Number analyzed (Participants) | 63 | 71
ms | 793.71 (101.74) | 808.20 (100.63)

ADVERSE EVENTS:
Time Frame: During a <2 hour laboratory session.
Description: As the study was short (< 2 hours), did not involve any medical procedures, and recruited healthy couples with no major chronic disease, no serious adverse events were expected to occur. Previous research using similar procedures of stimulation (of similar intensity) also suggests that adverse events are unlikely. At most, mild forms of adverse events could occur in terms of physical irritation from stimulation and were monitored. Mortality/serious adverse events were not monitored/assessed.
Arm/Group | Active tVNS | Sham tVNS
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/160 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-03-01): https://cdn.clinicaltrials.gov/large-docs/13/NCT05899413/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05899413/ICF_001.pdf